CLINICAL TRIAL: NCT01624558
Title: Effectiveness of Carbon Filters to Reduce the Anesthetic Gas Concentration in an Anesthetized Patient
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Measurement device not performing to standard in study environment
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Robert Greenberg, MD, Associate Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00049358
Record Dates: First submitted 2012-06-11; First posted 2012-06-20 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Malignant Hyperthermia
Keywords: malignant hyperthermia
MeSH Terms: conditions — Malignant Hyperthermia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (filter in circuit) (Experimental): After baseline use of volatile anesthetic, this group will have carbon filter placed in-line.
  Interventions: Device: In-line Carbon filter (Vapor-Clean)
- No Intervention Control (No Intervention): After baseline use of volatile anesthetic, this group will NOT have carbon filter placed in-line.

INTERVENTIONS:
Device: In-line Carbon filter (Vapor-Clean) — Carbon filter placed in anesthesia breathing circuit.
  Other Names: Vapor-Clean Brand Carbon Filter (Dynasthetics, LLC)
  Arms: Treatment (filter in circuit)

SUMMARY:
Malignant hyperthermia is a potentially fatal inherited disorder triggered by exposure to volatile anesthetic gases, most commonly recognized in children during anesthesia. Carbon filters have been used to scavenge various gases. A new carbon filter (Vapor Clean, Dynasthetics, LLC, Salt Lake City, Utah) with a 510(k) clearance specifically for scavenging anesthetic gases is being marketed, though the filter itself has never been studied in vivo. Bench studies conducted by the manufacturer of the product demonstrate it is extremely effective in reducing the volatile gas output from an anesthesia machine within 2 minutes. This pilot study will measure the effect on volatile gas concentration in non-malignant hyperthermia susceptible patients. Twelve (12) patients will undergo standard anesthetic induction using inhalational anesthetic (Sevoflurane®) and maintained on 3% for 30 minutes to attain steady state concentrations.1 At that time, a total intravenous anesthetic technique will be started and maintained throughout the case. Simultaneously a Vapor Clean filterset will be placed in the breathing circuit (inspiratory and expiratory limbs). Volatile gas concentration will be measured and recorded. This research will determine the feasibility of using this carbon filter to quickly reduce the breathing circuit gas concentration of volatile anesthetic in the clinical setting. This is fundamental in establishing this as a key life saving measure in eliminating the stimulus in a malignant hyperthermia event.

DETAILED DESCRIPTION:
see above.

ELIGIBILITY:
Inclusion Criteria:

* healthy ASA PS I or II children 2 years to 16 years old
* having general anesthesia for approximately 1 hour or more

Exclusion Criteria:

* malignant hyperthermia susceptible patients (personal or family history)
* patients with known neuromuscular disorders at high risk of malignant hyperthermia (e.g., muscular dystrophy)
* egg or soy allergy
* patient or parent refusal
* pregnant patients

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Time to reduce Concentration of Volatile Anesthetic to <5ppm | every two minutes after filter applied until concentration is <5ppm or 30 minutes
  At regular intervals (2 minutes) after application of the filters, the concentration of the volatile anesthetic will be measured. Primary outcome value will be the time to reduce breathing circuit volatile anesthetic concentration to <5ppm. If at 30 min the concentration is not <5ppm, then collection will be stopped.

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Greenberg, MD, Principal Investigator — Johns Hopkins University